CLINICAL TRIAL: NCT05409950
Title: Evaluation of Socket Shield Technique With Immediate Implant Placement in the Esthetic Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Russian University (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR-1
Record Dates: First submitted 2022-05-24; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Alveolar Bone Resorption
Keywords: Immediate implants, sockets shield technique, esthetic zone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group: implants were inserted using socket shield technique at the esthetic zone (Active Comparator)
  Interventions: Procedure: Immediate implant placement using socket shield technique
- Control group: implants were inserted using conventional immediate technique (No Intervention)

INTERVENTIONS:
Procedure: Immediate implant placement using socket shield technique — Evaluation of socket shield technique with immediate implant placement at the esthetic zone in comparison with the conventional immediate implant placement
  Arms: Study group: implants were inserted using socket shield technique at the esthetic zone

SUMMARY:
The study was conducted on 20 immediate implant placement sites in the anterior maxillary region. In the study group, 10 implants were inserted using socket shield technique, while in control group, 10 implants were inserted using conventional immediate placement technique. All patients received immediate and 6 months post-operative CBCT to assess horizontal bone loss, vertical bone loss, and measurement of bone density. Implant stability quotients (ISQs) was measured immediately, 1st, 3rd and 6 months post-operatively.

DETAILED DESCRIPTION:
Unrestorable tooth extraction with immediate implant placement is considered one of the best treatment options in restoring the esthetics and function. Extraction socket resorption is considered a challenging procedure when it involves the esthetics zone. The preservation of the entire attachment apparatus for complete preservation of the alveolar ridge makes socket shield technique a promising procedure that helps to maintain anatomy, esthetics and function. Socket shield technique, eliminate the negative consequences of bone resorption of the buccal plate of bone; leading to maintaining hard and soft tissue contours and provides a perfect pleasing esthetic result with good function. It is a highly promising technique in terms of maintaining pink and white esthetics through preservation of the interdental papilla during preparation of the interdental socket shield. It is considered a minimally invasive surgical procedure and offers the advantages of immediate implant placement.

ELIGIBILITY:
Inclusion Criteria:

1. Endodontic or non-endodontic treated un-restorable remaining root/ tooth related to maxillary anterior teeth.
2. Healthy adult patients > 20 years old (ASAI, II) .
3. Adequate oral hygiene.
4. Intact periodontal tissues.

Exclusion Criteria:

1. Periapical or periodontal active infection involving the teeth/root to be extracted (as excluded by radiographic examination).
2. Medically compromised patients (ASA III, IV, V).
3. Patients receiving chemotherapy or radiotherapy.
4. Heavy smokers,alcohol or drug abuse.
5. Patients with parafunctional habits such as bruxism, clenching, excessive gum chewing, lip or fingernail biting.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Implant stability | immediate postoperative
  Using osstell
Implant stability | one month post-operative
  Using osstell
Implant stability | three month post-operative
  Using osstell
Implant stability | six month post-operative
  Using osstell
Horizontal gap | immediate postoperative
  Using cone-beam computed tomography
Horizontal gap | six month post-operative
  Using cone-beam computed tomography
Vertical bone loss | immediate postoperative
  Using cone-beam computed tomography
Vertical bone loss | six month post-operative
  Using cone-beam computed tomography
Bone density | immediate postoperative
  Using cone-beam computed tomography
Bone density | six month post-operative
  Using cone-beam computed tomography
peri-implant probing depth | immediate postoperative
  using periodontal probe
peri-implant probing depth | one month post-operative
  using periodontal probe
peri-implant probing depth | three month post-operative
  using periodontal probe
peri-implant probing depth | six month post-operative
  using periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Suez canal university, Ismailia, Egypt